### 1.0 Title Page

### **Statistical Analysis Plan**

### **Study M13-596**

A Single-Arm, Open-Label, Multicenter Study to Evaluate the Safety and Efficacy of ABT-493/ABT-530 in Adult Post-Liver or Post-Renal Transplant Recipients with Chronic Hepatitis C Virus Genotype 1 – 6 Infection (MAGELLAN-2)

Date: 27 October 2016

| 2.0 | Table of Contents | |
|---|---|---|
| 1.0 | Title Page | 1 |
| 2.0 | Table of Contents | |
| 3.0 | Introduction | 5 |
| 4.0 | Study Objectives, Design and Procedures | 5 |
| 4.1 | Objectives | 5 |
| 4.2 | Design Diagram | 6 |
| 4.3 | Sample Size | 6 |
| 4.3.1 | Justification of Non-Inferiority Margin for SVR <sub>12</sub> | 7 |
| 4.4 | Primary Analyses | 8 |
| 5.0 | Analysis Populations | 8 |
| 5.1 | Definition for Analysis Populations | 8 |
| 5.1.1 | Intention-to-Treat (ITT) Population | 8 |
| 5.1.2 | Modified Intention-to-Treat (mITT) Populations | 8 |
| 5.1.3 | Safety Population | 9 |
| 5.2 | Variables Used for Stratification of Randomization | 9 |
| 6.0 | Analysis Conventions | 9 |
| 6.1 | Definition of Baseline and End of Treatment Assessment | 9 |
| 6.1.1 | Baseline | 9 |
| 6.1.2 | Study Days | 10 |
| 6.2 | Definition of Analysis Windows | 10 |
| 6.3 | Missing Data Imputation | 13 |
| 7.0 | Demographics, Baseline Characteristics, Medical History, and Other Medications | 14 |
| 7.1 | Demographic and Baseline Characteristics | |
| 7.2 | Medical History | |
| 7.3 | Prior, Concomitant and Post-Treatment Medications | 20 |
| 8.0 | Patient Disposition | |
| 8.1 | Disposition of Safety Population | |
| 9.0 | Study Drug Exposure and Compliance | |
| 9.1 | Exposure | |
| 9.2 | Compliance | 22 |

| 10.0 | Efficacy Analysis | 23 |
|--------|---------------------------------------------------------------|----|
| 10.1 | General Considerations | |
| 10.2 | Handling of Multiplicity | 27 |
| 10.3 | Primary Efficacy Analysis | 27 |
| 10.4 | Secondary Efficacy Analyses | 27 |
| 10.5 | Sensitivity Analyses for SVR | 28 |
| 10.5.1 | Imputation Approaches | 28 |
| 10.6 | Efficacy Subgroup Analysis | 29 |
| 10.7 | Additional Efficacy Analyses | 30 |
| 10.8 | Resistance Analyses | 32 |
| 10.8.1 | Presence of Baseline Resistance-Associated Variants | 37 |
| 10.9 | Patient Reported Outcomes | 39 |
| 11.0 | Safety Analysis | 40 |
| 11.1 | General Considerations | 40 |
| 11.2 | Analysis of Adverse Events | 40 |
| 11.2.1 | Treatment-Emergent Adverse Events | 40 |
| 11.2.2 | Tabulations of Treatment-Emergent Adverse Events | 41 |
| 11.2.3 | Listing of Adverse Events | 44 |
| 11.3 | Analysis of Laboratory Data | 44 |
| 11.3.1 | Variables and Criteria Defining Abnormality | 44 |
| 11.3.2 | Statistical Methods | 45 |
| 11.4 | Analysis of Vital Signs and Weight | 47 |
| 11.4.1 | Variables and Criteria Defining Abnormality | 47 |
| 11.4.2 | Statistical Methods | 48 |
| 12.0 | Summary of Changes | 49 |
| 12.1 | Summary of Changes Between the Latest Version of Protocol and | |
| 12.0 | SAP | |
| 13.0 | References | 4Y |



## **List of Tables**

| Table 1. | Analysis Time Windows for HCV RNA, Resistance Endpoints,<br>Laboratory, Vital Sign Measurements and PRO Instruments<br>(Treatment Period) | 11 |
|---|---|---|
| Table 2. | Analysis Time Windows for HCV RNA and Resistance Endpoints (Post-Treatment Period) | 12 |
| Table 3. | Laboratory Data, Vital Sign and PRO Instruments Visit Windows (Post-Treatment Period) | 13 |
| Table 4. | Baseline Fibrosis Stage | 18 |
| Table 5. | Medical History eCRF | 19 |
| Table 6. | List of Genotype-Specific Signature Amino Acid Positions and a<br>Key Subset of Amino Acid Positions | 33 |
| Table 7. | Resistance-Associated Variants by DAA Target and HCV Genotype | 38 |
| Table 8. | Definitions of Toxicity Grades 1, 2, 3, and 4 for Laboratory Values | |
| Table 9. | Criteria for Potentially Clinically Significant Vital Sign Values | 48 |
| List of Fi | igures | |
| Figure 1 | Study Schematic | e |



### 3.0 Introduction

This statistical analysis plan (SAP) describes the statistical analyses to be completed by the AbbVie Statistics and Statistical Programming Departments, or designee, for Study M13-596. Study M13-596 examines the safety and efficacy of 12 weeks of treatment with the ABT-493/ABT-530 combination regimen in adults with HCV GT1 – 6 infection who are DAA-naïve and post primary orthotopic liver transplant or renal transplant.

This SAP (Version 1.0) provides details to further elaborate the statistical methods outlined in Clinical Study Protocol M13-596 Amendment 1 dated 26 May 2016 and describes analysis conventions to guide the statistical programming. Analyses will be performed using SAS® Version 9.3 (SAS Institute, Inc., Cary, NC) or later under the UNIX operating system.

### 4.0 Study Objectives, Design and Procedures

### 4.1 Objectives

The primary objectives of this study are to compare the 12-week sustained virologic response,  $SVR_{12}$  (HCV RNA < LLOQ 12 weeks following therapy) of 12 weeks of treatment with the ABT-493/ABT-530 combination regimen in adults with HCV GT1 – 6 infection and post primary orthotopic liver transplant or renal transplant to a pre-defined threshold, based on the historical  $SVR_{12}$  rates for the current standard of care regimens (sofosbuvir/ledipasvir plus ribavirin or sofosbuvir plus daclatasvir plus RBV) and to assess the safety of treatment with the ABT-493/ABT-530 combination regimen for 12 weeks in adults with HCV GT1 – 6 infection and post primary orthotopic liver transplant or renal transplant.

The secondary objectives are to assess the percentage of subjects with on-treatment virologic failure, and the percentage of subjects with post-treatment relapse.

The pharmacokinetics and the emergence and persistence of viral variants for this treatment regimen also will be assessed.

### 4.2 Design Diagram

This is a Phase 3, single arm, open-label, multicenter study evaluating the safety and efficacy of ABT-493/ABT-530 for 12 weeks, in GT1 – 6 HCV-infected non-cirrhotic (F0-F3) subjects who have received a primary orthotopic liver or renal transplant who are either HCV treatment-naïve or prior treatment-experienced with IFN or pegIFN with or without RBV or sofosbuvir with RBV with or without pegIFN (except GT3-infected subjects who must be treatment-naïve).

This study consists of a Treatment Period and a Post-Treatment (PT) Period.

The study is designed to enroll approximately 90 subjects to meet scientific and regulatory objectives without enrolling an undue number of subjects in alignment with scientific and ethical considerations.

Figure 1. Study Schematic



#### 4.3 Sample Size

It is planned to enroll approximately 90 subjects with a minimum of 15 post-renal transplant subjects and a maximum of approximately 50 subjects with HCV genotype 1 infection in this study. The primary efficacy endpoint of SVR<sub>12</sub> will be assessed for the ITT population. For the primary efficacy endpoint of SVR<sub>12</sub>, with a sample size of 90 subjects and assuming that 96% of the subjects will achieve SVR<sub>12</sub>, this study has



greater than 90% power to show non-inferiority to the historical SVR<sub>12</sub> rate of 94% (based on the lower bound of a normal approximation of a single binomial proportion confidence interval being above a threshold of 86%) using a one-sample test for superiority using EAST 6.3.

| The 86% threshold was established by applying an 8% non-inferiority margin to the |
|---|
| historical SVR <sub>12</sub> rate of 94% |

No adjustment for dropouts is applicable because subjects who do not have data at Post-Treatment Week 12 (after imputing) are counted as failures for  $SVR_{12}$ .

### 4.3.1 Justification of Non-Inferiority Margin for SVR<sub>12</sub>

The 8% non-inferiority margin is based on the paucity of data in non-GT1 liver transplant recipients and renal transplant recipients regardless of genotype and the potential benefit of a RBV-free regimen.

- Most data published on the post-transplant population to date, including the studies that were used to establish the historical control rate for this study, are in GT1 subjects who have received a liver transplant.
- The current standard-of-care regimens used for historical comparison all include RBV. Given the ABT-493/ABT-530 regimen is RBV-sparing, a slightly wider non-inferiority margin compared to the margin used in other AbbVie Phase 3 studies with ABT-494/ABT-530 was considered, as a small decrement in efficacy may be outweighed by an improvement in safety offered with the avoidance of RBV in a patient population more susceptible to RBV related toxicity.



### 4.4 Primary Analyses

The primary analysis will occur after all subjects have completed the PT Week 12 Visit or prematurely discontinued the study. For the primary analysis, data will be locked after performing data cleaning. Results from the primary analysis (e.g., SVR<sub>12</sub> data) will be described in the primary clinical study report (CSR) that is planned to be included as part of submissions to regulatory agencies to support possible labeling changes.

The final analysis will be conducted when all subjects enrolled in the study have completed the 24 week post-treatment visit or prematurely discontinued from the study. Data after the primary analysis will be added to a new version of the database which will be cleaned and locked at the end of the study and included in the final CSR.

### 5.0 Analysis Populations

### 5.1 Definition for Analysis Populations

### 5.1.1 Intention-to-Treat (ITT) Population

All enrolled subjects who receive at least one dose of study drug will be included in the ITT population. Efficacy analyses will be performed on the ITT population.

### 5.1.2 Modified Intention-to-Treat (mITT) Populations

Sensitivity analyses of SVR<sub>12</sub> as described in Section 10.5, when applicable, will be performed on the ITT population modified to exclude subjects not of an eligible genotype (e.g., subjects of multiple/mixed genotypes or treatment-experienced subjects who were determined to be GT3 according to LiPA, Sanger or phylogenetic analyses as described in Section 10.8 under HCV Genotype/Subtype) (mITT-GT), and on the mITT-GT population further modified to exclude subjects who did not achieve SVR<sub>12</sub> for reasons other than virologic failure (mITT-GT-VF).



### 5.1.3 Safety Population

All subjects who receive at least one dose of study drug will be included in the safety population. Safety and demographic analyses will be performed on the safety population.

### 5.2 Variables Used for Stratification of Randomization

This study is not randomized. Eligible subjects will be enrolled into a single arm.

### 6.0 Analysis Conventions

#### 6.1 Definition of Baseline and End of Treatment Assessment

#### 6.1.1 Baseline

The baseline value refers to the last non-missing measurement collected before the first dose of study drug is received. The protocol specifies that all Day 1 assessments (other than optional intensive PK samples) are to be performed prior to administering the first dose of study drug. Therefore, all Day 1 assessments for which time is not collected will be assumed to be pre-dose and the baseline value will be the last non-missing measurement collected on or before the first day of study drug administration.

All Day 1 assessments with time available must be before the time of first dose to be considered baseline and the last non-missing measurement collected before the date and time of the first dose of study drug will be considered the baseline value. If multiple measurements that are prior to dosing are recorded on the same date and with the same time or if time is not available, then the average of these measurements will be considered the baseline value. The same baseline value will be used for analyses of the Treatment and Post-Treatment Periods.

Safety assessments that are related to a serious adverse event that occurred on the first dose day are excluded when applying this algorithm.



**ABT-493/ABT-530** 

M13-596 – Statistical Analysis Plan Version 1.0 – 27 October 2016

#### 6.1.2 **Study Days**

Study days are calculated for each time point relative to the first dose of study drug. Study days are negative values when the time point of interest is prior to the first study drug dose day. Study days are positive values when the time point of interest is after the first study drug dose day. There is no Study Day 0. Study Day 1 is the day of the first dose of study drug.

### Study Drug End Days (Days Relative to the Last Dose of Study Drug)

Study drug end days are calculated for each time point relative to the last dose of study drug. The last day of study drug dosing is defined as Study Drug End Day 0. Days before it have negative study drug end days and days after it have positive study drug end days.

#### **Final Treatment Value**

The final treatment value is defined as the last non-missing measurement collected after Study Day 1 and on or before Study Drug End Day 2.

#### **Final Post-Treatment Value**

The final post-treatment value for each subject is the last non-missing measurement collected after Study Drug End Day 2 and on or before Study Drug End Day 999.

#### 6.2 **Definition of Analysis Windows**

For efficacy analyses of HCV RNA and resistance, the time windows specified in Table 1 and Table 2 describe how efficacy data are assigned to protocol-specified time points during the Treatment and PT Periods, respectively. All time points and corresponding time windows are defined based on the date/time of blood sample collection.

For laboratory data vital signs and PRO measurements, the time windows specified in Table 1 and Table 3 describes how data are assigned to protocol specified time points.



If more than one assessment is included in a time window, the assessment closest (except in analyses of SVR) to the nominal time will be used. If there are two observations equally distant to the nominal time, the latest one will be used in analyses. For analyses of SVR (e.g., SVR<sub>12</sub>), the last value in the window will be used.

If multiple measurements are made on the same day for a safety laboratory parameter or a vital sign parameter, the average of the values will be used to calculate descriptive statistics and in analyses of the mean change from baseline. For summaries of shifts from baseline and potentially clinically significant values, multiple values on the same day will not be averaged; all values will be considered for these analyses.

Table 1. Analysis Time Windows for HCV RNA, Resistance Endpoints, Laboratory, Vital Sign Measurements and PRO Instruments (Treatment Period)

| Scheduled Visit | Nominal Day (Study Day) | Time Window (Study Day Range) |
|---|---|---|
| Day 1/Baseline <sup>a</sup> | 1 | ≤ 1 <sup>a</sup> |
| Day 3 | 3 | 2 to 5 |
| Week 1 | 7 | 6 to 8 |
| Day 10 | 10 | 9 to 12 |
| Week 2 | 14 | 13 to 21 |
| Week 4 | 28 | 22 to 42 |
| Week 6 | 42 | 43 to 49 |
| Week 8 | 56 | 50 to 70 |
| Week 12 | 84 | 71 to 98 |
| Final Treatment Visit <sup>b</sup> | 2 to $\leq$ 2 days after | last dose of study drug |

Day of first dose of study drug.

Note: Data must also have Study Drug End Day  $\leq 2$  for all windows. The result closest to the scheduled time point will be used. PRO instruments are collected at Day 1 and End of Treatment Visit (Week 12) only.

b. The last value within the window will be used to define the Final Treatment Visit value. The upper bound of this Final window is Study Drug End Day  $\leq 2$ .



Table 2. Analysis Time Windows for HCV RNA and Resistance Endpoints (Post-Treatment Period)

| Scheduled Visit <sup>a</sup> | Nominal Day<br>(Study Drug End Day) | Time Window<br>(Study Drug End Day Range) |
|---|---|---|
| Post-Treatment Week 2 | 14 | 3 to 21 |
| Post-Treatment Week 4 | 28 | 22 to 42 |
| Post-Treatment Week 8 | 56 | 43 to 70 |
| Post-Treatment Week 12 | 84 | 71 to 126 |
| Post-Treatment Week 24 | 168 | 127 to 999 |
| SVR <sub>4</sub> <sup>b</sup> | 28 | 3 to 56 |
| SVR <sub>12</sub> <sup>b</sup> | 84 | 57 to 126 |
| SVR <sub>24</sub> <sup>b</sup> | 168 | 127 to 210 |

a. Post-Treatment Visits are applicable for subjects who received at least one dose of study drug.

Note: The result closest to the scheduled time point will be used, except for  $SVR_4$ ,  $SVR_{12}$ , and  $SVR_{24}$ . Data must also have Study Drug End Day > 2 for all windows. Study Drug End Day 0 is defined as the day of the last dose of study drug.

b. For SVR windows, the last value in the window will be used.



Table 3. Laboratory Data, Vital Sign and PRO Instruments Visit Windows (Post-Treatment Period)

| | Nominal Day | Time Window<br>(Study Drug End Days Range) |
|---|---|---|
| <b>Scheduled Time</b> | (Study Drug End Day) | Vital Sign |
| Post-Treatment Day 3 | 3 | 3 to 5 |
| Post-Treatment Week 1 | 7 | 6 to 10 |
| Post-Treatment Week 2 | 14 | 11 to 21 |
| Post-Treatment Week 4 | 28 | 22 to 42 |
| Post-Treatment Week 8 | 56 | 43 to 70 |
| Post-Treatment Week 12 | 84 | 71 to 126 |
| Post-Treatment Week 24 | 168 | 127 to 999 |
| Final Post-Treatment Visit <sup>a</sup> | > 2 days af | ter last dose of study drug |

a. The last value within the Post-Treatment Period window will be used to define the final post-treatment value. The lower bound of this Final window is Study Drug End Day 3.

Note: The result closest to the scheduled time point will be used. Data must also have Study Drug End Day > 2. Vital signs are collected at every PT visit; hematology, chemistry, urinalysis, and coagulation panels are collected at every PT visit except PTW8 and PTW12. PRO instruments are collected at PTW12 and PTW24 (or PTDC) only.

#### 6.3 Missing Data Imputation

### **Missing Data Imputation for SVR**

HCV RNA values will be selected for analysis based on the analysis windows defined in Section 6.2.

For analyses of SVR, subjects missing visit values will have backward imputation applied, if possible. For backward imputation, if the nearest HCV RNA value after the SVR window is unquantifiable or undetectable, then it will be used to impute the HCV RNA value in the SVR window. If a subject is missing an HCV RNA value within the appropriate SVR window after performing backward imputation, then this value will be imputed with an HCV RNA value from a local laboratory if present; otherwise, the HCV RNA value will be missing. Subjects with missing HCV RNA data in the analysis window, after imputations, will be imputed as a failure.



abbvie ABT-493/ABT-530

M13-596 – Statistical Analysis Plan Version 1.0 – 27 October 2016

Regardless of the imputation method described above, if a subject starts another treatment for HCV, then all HCV RNA values for this subject measured on or after the start date of the new HCV treatment will be excluded from analyses. The subject will be considered a failure for summaries of viral response at all time points after the start of the new HCV treatment.

#### Missing Data Imputation for Virologic Failure

If HCV RNA values from the central laboratory are missing but a local laboratory value is present in the appropriate time period, then the local laboratory value will be used to assess post-treatment relapse and on-treatment virologic failure.

#### Missing Data Imputation for PRO Questionnaires

The handling of missing data for patient reported outcomes (PROs) will be as follows. If a respondent answers at least 50% of the items in a multi-item scale of the SF-36v2, the missing items will be imputed with the average score of the answered items in the same scale. In cases where the respondent did not answer at least 50% of the items, the score for that domain will be considered missing. The Mental and Physical Component Summary measures will not be computed if any domain is missing. The missing items of the FSS questionnaire will be imputed with the average score of the answered items as long as more than 50% of the items on the FSS are answered. For EQ-5D-3L index and VAS scores, no imputation will be performed for missing items.

#### 7.0 **Demographics, Baseline Characteristics, Medical** History, and Other Medications

Demographics and baseline characteristics will be summarized on the safety population overall and by type of transplant (liver or kidney).

The safety population will be used to summarize medical history and previous, concomitant, and post-treatment medications.



### 7.1 Demographic and Baseline Characteristics

Categorical demographic and baseline characteristic variables will be summarized with the number and percentage of subjects. Continuous variables will be summarized with descriptive statistics (number of non-missing observations, mean, standard deviation, median, maximum and minimum).

Continuous demographic variables include age, weight, height, and body mass index (BMI). Categorical demographic variables include sex, race, black race (black or non-black), ethnicity, age category (< 65 or  $\ge$  65 years; < 75 or  $\ge$  75 years), BMI category (< 30, or  $\ge$  30 kg/m<sup>2</sup>), country, and geographic region (North America, Europe, or rest of world [ROW]).

When defining geographic region, sites in the United States, Canada, and Puerto Rico will be grouped under North America; sites in Italy, Spain, and the United Kingdom will be grouped under Europe; sites in Australia, New Zealand, and Taiwan will be grouped together as ROW).

Continuous baseline characteristics include baseline  $log_{10}$  HCV RNA level, homeostasis model of assessment – insulin resistance (HOMA-IR), creatinine clearance, eGFR, platelet count, albumin, GGT, LDL, HDL, APRI, FIB-4, AST, ALT, total, direct, indirect bilirubin, and time since transplantation (months).

Categorical baseline characteristics include:

- HCV genotype (1, 2, 3, 4, 5, or 6) and available subtype (as determined by the central laboratory);
- Prior HCV treatment history (treatment-naïve or treatment-experienced);
  - For treatment-experienced subjects, type of previous regimen (IFN-, SOF-based, or other);
  - For treatment experienced subjects, type of non-response to previous treatment (on-treatment non-responder or breakthrough, post-treatment relapse, or unknown/other);



- For treatment-experienced subjects, occurrence of prior HCV treatment relative to renal or liver transplant (pre-transplant or post-transplant);
- Prior HCV DAA treatment history:
  - DAA-naïve (i.e., treatment naïve or treatment-experienced with IFN or pegIFN with or without RBV);
  - SOF-experienced (i.e., treatment-experienced with sofosbuvir with RBV with or without pegIFN);
  - Other DAA-experienced (i.e., treatment-experienced with DAA drugs other than sofosbuvir);
- IL28B genotype (CC, CT, or TT; CC or non-CC);
- Baseline HCV RNA level (< 1,000,000 or  $\geq$  1,000,000 IU/mL; < 6,000,000 or  $\geq$  6,000,000 IU/mL);
- Baseline creatinine clearance ( $< 60, \ge 60 \text{ to } < 90, \ge 90 \text{ mL/min}$ );
- Baseline eGFR ( $< 60, \ge 60 \text{ to } < 90, \ge 90 \text{ mL/min/1.73 m}^2$ );
- Baseline fibrosis stage (equivalent to Metavir F0 F1, F2, F3, or F4 [if applicable]);
- Baseline platelet count ( $< 90 \text{ or } \ge 90 \times 10^9/\text{L}$ );
- Baseline albumin ( $< 35 \text{ or } \ge 35 \text{ g/L}$ );
- History of diabetes (yes/no);
- History of bleeding disorders (yes/no);
- History of depression or bipolar disorder (yes/no);
- History of cardiovascular disease (yes/no);
- Type of transplant (liver or kidney),
  - For renal transplant subjects, prior dialysis type (hemodialysis, peritoneal dialysis, other, or not done);
- Donor type (living or deceased);
- Immunosuppressant medication (Tacrolimus, Cyclosporine, other);
- Injection drug user (yes, within last 12 months; yes, more than 12 months ago; or no);
- Subject on stable opiate substitution (yes/no);



- Tobacco use (user, ex-user, or non-user);
- Alcohol use (drinker, ex-drinker, or non-drinker);
- Concomitant use of Proton Pump Inhibitors (PPIs).

Summaries of baseline resistance are described in Section 10.8.

Any concomitant medication coded to the WHO Drug Dictionary ATC code of A02BC will be counted as a PPI.

If the IL28B genotype result is not available from a sample collected on Day 1, then a result available from a sample collected at any time during the study will be used to summarize IL28B genotype. IL28B rs12979860 will be resulted as C/C, C/T, or T/T by the central laboratory.

HOMA-IR is defined as fasting glucose (mmol/L)  $\times$  fasting insulin ( $\mu$ IU/mL)  $\div$  22.5. Subjects who do not have concurrent fasting glucose and fasting insulin values at baseline will be excluded from the summary of baseline HOMA-IR.

Baseline fibrosis stage is defined for subjects with non-missing liver biopsy scores, FibroScan scores, or FibroTest scores. Only one score will be used to categorize each subject even if a subject has more than one score recorded. If a biopsy score is present, then it will be used to categorize the subject, regardless of the FibroScan/FibroTest score. Similarly, if a FibroScan score is present along with a FibroTest score, then the FibroScan score will be used to categorize the subject. If biopsy and FibroScan scores are not present and more than one FibroTest result is available, then the baseline FibroTest result (i.e., last non-missing FibroTest result on or before Day 1) will be used to categorize the subject. Subjects will be categorized as F0 – F1, F2, F3, or F4 according to Table 4.

All subjects will be categorized as not having cirrhosis (cirrhosis = no) since this study excludes subjects with cirrhosis.

Table 4.Baseline Fibrosis Stage

| Baseline Fibrosis<br>Stage, Metavir<br>Equivalents | Liver Biopsy Metavir, Batts<br>Ludwig, Knodell, IASL,<br>Scheuer, or Laennec Score | Liver Biopsy<br>Ishak Score | FibroScan<br>(kPa) | FibroTest* |
|---|---|---|---|---|
| F0 – F1 | 0 or 1 | 0, 1, or 2 | < 8.8 | ≤ 0.48 |
| F2 | 2 | 3 | $\geq$ 8.8 to $\leq$ 9.6 | 0.49 to 0.58 |
| F3 | 3 | 4 | $\geq$ 9.6 to < 12.5 | 0.59 to 0.74 |
| F4 | 4 | ≥ 5 | ≥ 12.5 | $\geq 0.75$ |

<sup>\*</sup> APRI will not be used to derive Baseline Fibrosis Stage. However, per inclusion/exclusion criteria, subjects need to have concordant FibroTest and APRI scores in order to determine eligibility.

Immunosuppressant medications (i.e., Cyclosporine, Sirolimus, Everolimus and Tacrolimus) are captured on the "Immunosuppression Regimen Dosing Diary" eCRF. Other immunosuppressant medications are captured on the "Concomitant Medications and Supplements" eCRF.

Baseline APRI and FIB-4 are defined as the equations below. Subjects who do not have concurrent AST and platelet values at baseline will be excluded from the summary of baseline APRI. Age is defined in years at baseline. Subjects who do not have concurrent baseline values of AST, ALT, and platelet count or subjects who are missing age will be excluded from the summary of FIB-4.

$$APRI = \frac{\frac{AST \text{ Level (U/L)}}{AST \text{ (Upper Limit of Normal)(U/L)}}}{\text{Platelet Count (10}^{9}/\text{L)}} \times 100$$

$$FIB-4 = \frac{Age (years) \times AST Level (U/L)}{Platelet Count (10^9/L) \times \sqrt{ALT (U/L)}}$$

Histories of diabetes, bleeding disorders, depression or bipolar disorder, and cardiovascular disease will be based on the Medical History (MH) eCRF, as defined in Table 5.



Table 5. Medical History eCRF

| | Medical History eCRF | |
|---|---|---|
| Subgroup | Body System | Condition/Diagnosis |
| Diabetes | Metabolic | Diabetes mellitus |
| Bleeding disorders | Blood | Clotting/bleeding problems Factor deficiency Hemophilia Von Willebrand disease |
| Depression or bipolar disorder | Neurologic and Psychiatric<br>System | Bipolar disorder<br>Depression |
| Cardiovascular disease | Cardiovascular | Angina Cardiac arrhythmia Cardiovascular disease Congenital heart disease Congestive heart failure Coronary artery disease Hypertension Myocardial infarction Myocarditis Peripheral vascular disease-arterial Peripheral vascular disease-venous Valvular heart disease Vasculitis |

### 7.2 Medical History

Medical history data will be summarized and presented using body systems and conditions/diagnoses as captured on the eCRF. The body systems will be presented in alphabetical order and the conditions/diagnoses will be presented in alphabetical order within each body system. The number and percentage of subjects with a particular condition/diagnosis will be summarized. Subjects reporting more than one condition/diagnosis within a body system will be counted only once for that body system.



#### 7.3 Prior, Concomitant and Post-Treatment Medications

A prior medication is defined as any medication taken prior to the date of the first dose of study drug (ABT-493/ABT-530). A concomitant medication is defined as any medication that started prior to the date of the first dose of study drug and continued to be taken on or after the first dose of study drug or any medication that started on or after the date of the first dose of study drug, but not after the date of the last dose of study drug. A post-treatment medication for the treatment of HCV is defined as any medication taken on or after the last dose of study drug and entered as "Post-treatment HCV medications" on the eCRF.

The number and percentage of subjects taking prior medications, concomitant medications, and post-treatment HCV medications will be summarized by generic drug name based on the WHO Drug Dictionary. The prior HCV medications taken by the treatment experienced subjects will be summarized separately from other prior medications

The number and percentage of subjects taking concomitant immunosuppressant medications will be summarized separately from other concomitant medications.

The number and percentage of subjects with immunosuppressant medication dosage increase and decrease, respectively, at each post-baseline visit in the treatment period will be summarized by each immunosuppressant medication as captured on the "Immunosuppression Regimen Dosing Diary" eCRF (i.e., Cyclosporine, Sirolimus, Everolimus and Tacrolimus).

### 8.0 Patient Disposition

The number and percentage of subjects who screen failed for any reason, and for each screen fail reason, will be summarized for all subjects who screen failed.



### 8.1 Disposition of Safety Population

The number of subjects in each of the following categories will be summarized overall and by investigator.

- Subjects enrolled in this study;
- Subjects who took at least one dose of study drug;
- Subjects who completed study drug;
- Subjects who prematurely discontinued study drug;
- Subjects who completed the study;
- Subjects who prematurely discontinued from the study;
- Subjects ongoing in the Post-Treatment Period at the time of the primary analysis.

The number and percentage of subjects who discontinued study drug will be summarized by reason (all reasons) and by primary reason (per eCRF). Similar summaries will be provided for discontinuations from the study.

The number and percentage of subjects with reported study drug interruptions will be summarized.

Reasons for study drug interruptions will be presented in the CSR listings.

# 9.0 Study Drug Exposure and Compliance

#### 9.1 Exposure

The duration of exposure to study drug will be summarized for the safety population. Duration of exposure is defined for each subject as the last study drug dose date minus the first study drug dose date plus 1 day.

Descriptive statistics (mean, standard deviation, median, minimum, and maximum) will be presented for exposure during the treatment period.



Study drug duration will be summarized with frequencies and percentages using the following categories:

- 1 to 15 days
- 16 to 30 days
- 31 to 45 days
- 46 to 60 days
- 61 to 75 days
- 76 to 90 days
- > 90 days

In addition, the number and percentage of subjects with study drug duration of  $\geq$  77 days will be summarized.

### 9.2 Compliance

At each visit (starting with the Week 4 visit) during the Treatment Period, the total number of tablets dispensed and returned is recorded. The compliance for study drug (ABT-493/ABT-530) during the treatment period will be calculated as the percentage of tablets taken relative to the total tablets expected to be taken. The total number of tablets expected to be taken will be equal to the total number of tablets that should have been taken per the protocol for the duration that the subject was in the Treatment Period (date of last dose of study drug – date of first dose of study drug + 1). Study drug interruptions recorded on the eCRF will not be subtracted from the duration.

A subject is considered to be compliant if the percentage is between 80% and 120%. Compliance will be calculated for each subject and summarized with the mean, median, standard deviation, minimum, and maximum. The percentage of compliant subjects will be summarized for study drug, based on data as observed. An additional summary of the percentage of compliant subjects will be provided where subjects who are missing study drug accountability records will be imputed as non-compliant.



abbvie ABT-493/ABT-530

M13-596 – Statistical Analysis Plan Version 1.0 – 27 October 2016

#### 10.0 **Efficacy Analysis**

#### 10.1 **General Considerations**

#### **General Considerations**

All efficacy analyses will be performed on the ITT population, unless otherwise specified.

Missing data will be imputed as described in Section 6.3 for analyses of the HCV RNA endpoints of SVR.

Plasma HCV RNA levels will be determined for each sample collected by the central laboratory using the Roche COBAS® AmpliPrep/COBAS® TaqMan® HCV Quantitative Test, v2.0. The lower limit of detection (LLOD) and lower limit of quantification (LLOQ) for this assay (regardless of genotype) are both 15 IU/mL.

HCV RNA results that are detectable but not quantifiable are reported as "< 15 IU/ML HCV RNA DETECTED" and those that are undetectable are reported as "HCV RNA NOT DETECTED" in the database.

The notation "HCV RNA < LLOQ" is used to represent all HCV RNA values < 15 IU/mL, including values reported as "HCV RNA NOT DETECTED" or "< 15 IU/ML HCV RNA DETECTED." HCV RNA ≥ LLOQ are all quantifiable values of 15 IU/mL or greater.

#### **Definitions for Efficacy Endpoints**

A confirmed quantifiable value during treatment is defined as any two consecutive HCV RNA measurements  $\geq$  LLOQ (or 100 IU/mL for **Breakthrough**), either both during treatment or at the final treatment measurement and the next consecutive post-treatment measurement. A confirmed quantifiable post-treatment value is defined as any two consecutive post-treatment HCV RNA measurements  $\geq$  LLOQ.

**Breakthrough** = confirmed HCV RNA ≥ 100 IU/mL after HCV RNA < LLOQ during the Treatment Period; or confirmed increase from nadir in HCV RNA (two consecutive HCV RNA measurements  $> 1 \log_{10} IU/mL$  above nadir) at any time point during the Treatment Period. A single breakthrough value ( $\geq 100 \text{ IU/mL} \text{ or } > 1 \log_{10} \text{ above nadir}$ ) followed by lost to follow-up also will be considered a breakthrough (i.e., will not require confirmation).

**EOT failure** = HCV RNA \ge LLOQ at end of treatment with at least 6 weeks of treatment, where the HCV RNA value must be collected on or after Study Drug Day 36 and study drug duration  $\geq$  36 days.

**On-treatment virologic failure = Breakthrough or EOT failure.** 

 $SVR_4 = HCV RNA < LLOQ$  in the  $SVR_4$  window (4 weeks after the last actual dose of study drug) without any confirmed quantifiable (≥ LLOQ) post-treatment value before or during that SVR window.

 $SVR_{12} = HCV RNA < LLOQ$  in the  $SVR_{12}$  window (12 weeks after the last actual dose of study drug) without any confirmed quantifiable (≥ LLOQ) post-treatment value before or during that SVR window.

 $SVR_{24} = HCV RNA < LLOQ$  in the  $SVR_{24}$  window (24 weeks after the last actual dose of study drug) without any confirmed quantifiable (≥ LLOQ) post-treatment value before or during that SVR window.

**Relapse**<sub>12</sub> = confirmed HCV RNA  $\geq$  LLOQ between end of treatment and 12 weeks after last actual dose of study drug (up to and including the SVR<sub>12</sub> assessment time point) for a subject with HCV RNA < LLOQ at Final Treatment Visit who completed treatment (defined as study drug duration  $\geq 77$  days), excluding reinfection as described below.

**Relapse<sub>24</sub>** = confirmed HCV RNA  $\geq$  LLOQ within the SVR<sub>24</sub> window for a subject who achieved SVR<sub>12</sub> and has HCV RNA data available in the SVR<sub>24</sub> window, excluding reinfection.



**Relapse**<sub>overall</sub> = confirmed HCV RNA  $\geq$  LLOQ between end of treatment and up to and including the last HCV RNA measurement collected in the PT Period for a subject with HCV RNA  $\leq$  LLOQ at Final Treatment Visit who completed treatment (defined as study drug duration  $\geq$  77 days), excluding reinfection.

#### Virologic failure = On-treatment virologic failure or Relapse<sub>overall</sub>.

Only subjects who have at least one post-treatment HCV RNA value will be included in analyses of relapse. For the analysis of relapse, completion of treatment is defined as any subject with study drug duration of 77 days or greater. If the last available post-treatment value is  $\geq$  LLOQ, then the subject will be considered a relapse (i.e., will not require confirmation).

HCV reinfection is defined as confirmed HCV RNA ≥ LLOQ after the end of treatment in a subject who had HCV RNA < LLOQ at Final Treatment Visit, along with the post treatment detection of a different HCV genotype, subtype, or clade compared with baseline, as determined by phylogenetic analysis of the NS3 or NS5A, and/or NS5B gene sequences. Reinfection in the case of the same HCV subtype is defined as a clade switch, as indicated by the lack of clustering between the baseline and post-treatment sequences by phylogenetic analysis. If phylogenetic analysis is not possible due to technical difficulties, HCV reinfection may be determined with a confirmed HCV genotype or subgenotype switch by the Versant HCV Genotype Inno-LiPA Assay v2.0 or Sanger assay.

Post-treatment relapse is defined as described earlier (**Relapse**<sub>12</sub>, **Relapse**<sub>24</sub>, **Relapse**<sub>overall</sub>), and no genotype, subtype, or clade switch compared with baseline as determined by phylogenetic analysis of the NS3 or NS5A gene sequences. If phylogenetic analysis is not possible due to technical difficulties, the subject will be defined as having a post-treatment relapse unless an HCV genotype or subgenotype switch is confirmed by the Versant HCV Genotype Inno-LiPA Assay v2.0 or Sanger assay.



M13-596 – Statistical Analysis Plan Version 1.0 – 27 October 2016

### Reasons for SVR<sub>12</sub> Non-Response

Subjects who do not achieve SVR<sub>12</sub> (SVR<sub>12</sub> non-responders) will be categorized as having:

- 1. On-treatment virologic failure (see **On-treatment virologic failure** definition);
- 2. Relapse (defined according to the Relapse<sub>12</sub> definition for subjects who complete treatment);
- 3. Prematurely discontinued study drug with no on-treatment virologic failure (defined as any SVR<sub>12</sub> non-responder who prematurely discontinued study drug [study drug duration < 77 days] and did not meet the **On-treatment virologic** failure definition);
- 4. HCV reinfection (see definition described earlier);
- 5. Missing follow-up data in the SVR<sub>12</sub> window (defined as any subject who completed study drug without data in the SVR<sub>12</sub> window after applying the imputation rules and not meeting the definitions of [1], [2], [3], or [4]);
- 6. Other (defined as any SVR<sub>12</sub> non-responder not meeting the definitions of [1] - [5]).

### Reasons for SVR<sub>24</sub> Non-Response

Subjects who do not achieve SVR<sub>24</sub> (SVR<sub>24</sub> non-responders) will be categorized as having:

- 1. On-treatment virologic failure (see **On-treatment virologic failure** definition);
- 2. Relapse (defined according to the **Relapse**<sub>12</sub> definition for subjects who complete treatment);
- 3. Relapsed after achieving SVR<sub>12</sub> (see **Relapse<sub>24</sub>** definition);
- 4. Prematurely discontinued study drug with no on-treatment virologic failure (defined as any SVR<sub>24</sub> non-responder who prematurely discontinued study drug



[study drug duration < 77 days] and did not meet the **On-treatment virologic** failure, Relapse<sub>12</sub>, or Relapse<sub>24</sub> definitions);

- 5. HCV reinfection;
- 6. Missing follow-up data in the SVR<sub>24</sub> window (defined as any subject who completed study drug without data in the SVR<sub>24</sub> window after applying the imputation rules and not meeting the definitions of [1], [2], [3], [4], or [5]);
- 7. Other (defined as any SVR<sub>24</sub> non-responder not meeting the definitions of [1] [6]).

### 10.2 Handling of Multiplicity

No adjustment for multiple comparisons is used in this open-label single-arm study.

### 10.3 Primary Efficacy Analysis

The primary efficacy endpoint is  $SVR_{12}$  (HCV RNA < LLOQ 12 weeks after the last actual dose of study drug) in the ITT population. The number and percentage of subjects in the ITT population achieving  $SVR_{12}$  will be summarized with a two-sided 95% confidence interval, calculated using the normal approximation to the binomial distribution. If the  $SVR_{12}$  rate is 100%, then the Wilson's score method will be used to calculate the confidence interval.

The lower confidence bound of the 2-sided 95% CI (LCB) for the percentage of subjects achieving SVR<sub>12</sub> must exceed 86% to achieve non-inferiority to the standard of care.

### 10.4 Secondary Efficacy Analyses

Two secondary efficacy endpoints will be summarized:

• the percentage of subjects with on-treatment virologic failure (defined as **On-treatment virologic failure**);



• the percentage of subjects with post-treatment relapse (defined as **Relapse**<sub>12</sub>; subjects with reinfection will be summarized separately).

The number and percentage of subjects with on-treatment virologic failure and post-treatment relapse (**Relapse**<sub>12</sub>) will be summarized with two-sided 95% Wilson score intervals.

In addition, a summary of reasons for SVR<sub>12</sub> non-response (e.g., on-treatment virologic failure, relapse, other) will be provided.

### 10.5 Sensitivity Analyses for SVR

The following analysis approaches will be used as sensitivity analyses for the SVR<sub>12</sub> rate.

- A two-sided 95% confidence interval for the SVR<sub>12</sub> rate in the ITT population will be calculated using a Wilson score interval.
- The SVR<sub>12</sub> rate in the mITT-GT and mITT-GT-VF populations, as applicable, will be calculated, as well as the corresponding two-sided 95% confidence interval using a Wilson score interval and a Normal approximation to the binomial distribution.

Listings of subjects excluded from the mITT-GT and mITT-GT-VF populations will be provided, as applicable.

### 10.5.1 Imputation Approaches

In addition to imputing  $SVR_{12}$  as described in Section 6.3,  $SVR_{12}$  will be presented using the following other methods to impute missing HCV RNA values:

- imputing any missing HCV RNA values in the SVR<sub>12</sub> window by carrying forward the last non-missing (post-baseline) HCV RNA value prior to the SVR<sub>12</sub> window.
- impute as described in Section 6.3 but treat SVR<sub>12</sub> non-responders who were categorized as "prematurely discontinued study drug with no on-treatment



virologic failure" or "missing follow-up data in the SVR<sub>12</sub> window" as successes.

For each of these, the percentage of subjects with SVR<sub>12</sub> will be presented along with two-sided 95% Normal and Wilson score confidence intervals.

### 10.6 Efficacy Subgroup Analysis

The percentage of ITT subjects with SVR<sub>12</sub> will be calculated, as will the corresponding two-sided 95% Wilson score confidence intervals for the following subgroups:

- HCV genotype (1, 2, 3, 4, 5, or 6) and available subtype (as defined in Section 10.8);
- Prior HCV treatment history (treatment-naïve or treatment-experienced);
  - For treatment-experienced subjects, type of previous regimen (IFN- or SOF-based);
  - For treatment-experienced subjects, occurrence of prior HCV treatment relative to renal or liver transplant (pre-transplant or post-transplant);
- Type of organ transplant (liver or kidney);
- Type of immunosuppressant medications (Tacrolimus, Cyclosporine, or other);
- IL28B genotype (CC or non-CC);
- Sex (male or female);
- Age ( $< 65 \text{ or } \ge 65 \text{ years}$ ) and ( $< 75 \text{ or } \ge 75 \text{ years}$ );
- Race (White, Black/African-American, Asian, or other) and (black or non-black);
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino);
- Baseline BMI (< 30, or  $\ge 30 \text{ kg/m}^2$ );
- Baseline HCV RNA level ( $< 1,000,000 \text{ or } \ge 1,000,000 \text{ IU/mL}$ ) and ( $< 6,000,000,\text{ or } \ge 6,000,000 \text{ IU/mL}$ );
- Baseline fibrosis stage (equivalent to Metavir F0 F1, F2, F3, or F4 [if applicable]);
- Baseline platelet count ( $< 90 \text{ or } \ge 90 \times 10^9/\text{L}$ );



- Baseline albumin ( $< 35 \text{ or } \ge 35 \text{ g/L}$ );
- Baseline creatinine clearance ( $< 60, \ge 60 \text{ to } < 90, \ge 90 \text{ mL/min}$ );
- Baseline eGFR ( $< 60, \ge 60 \text{ to } < 90, \ge 90 \text{ mL/min/1.73 m}^2$ );
- Geographic region (North America, Europe, Rest of world);
- Country (as appropriate);
- History of diabetes (yes/no);
- Former injection drug user (yes, within last 12 months; yes, more than 12 months ago; or no);
- Subject on stable opiate substitution (yes/no);
- Presence of baseline resistance-associated variants (any NS3/4A variant [yes/no]; any NS5A variant [yes/no]; any NS3/4A and any NS5A variant [yes/no], any NS3/4A or any NS5A variant [yes/no]), and (NS3/4A variant only, NS5A variant only, both NS3/4A and NS5A, or none);
- Concomitant use of Proton Pump Inhibitors (PPIs) (yes/no).

The 2-sided 95% Wilson score confidence interval will be produced if there are at least 10 subjects in the subgroup.

For the subgroup analyses, the presence of baseline resistance-associated variants as listed above are defined in Section 10.8.1; this subgroup analysis will be performed in the mITT-GT-VF population.

### 10.7 Additional Efficacy Analyses

The following additional efficacy endpoints will be summarized:

- The percentage of subjects with HCV RNA < LLOQ at each post-baseline visit in the Treatment Period (using data as observed);
- The percentage of DAA-naïve subjects with on-treatment virologic failure;
- The percentage of DAA-naïve subjects with post-treatment relapse;
- The percentage of subjects with SVR<sub>4</sub>;
- The percentage of subjects with SVR<sub>24</sub>;



- The percentage of subjects who relapsed after achieving SVR<sub>12</sub> (**Relapse<sub>24</sub>**);
- The percentage of subjects with virologic failure through Post-Treatment Week 12 (i.e., the SVR<sub>12</sub> non-responders due to on-treatment virologic failure or Relapse<sub>12</sub>)

In the above analyses for SVR, virologic failure, and relapse, the percentage of subjects with a two-sided 95% Wilson score interval will be summarized. Imputations for missing data will be performed as described in Section 6.3 for analysis of SVR, where a missing response will be imputed as a failure after performing the described imputation. All other endpoints will be presented using data as observed.

A summary of the subjects who completed treatment and relapsed (defined as **Relapse**<sub>overall</sub>) will be prepared displaying the number of subjects relapsing overall and by SVR visit window (within the SVR<sub>4</sub>, SVR<sub>12</sub>, SVR<sub>24</sub> windows or after SVR<sub>24</sub> window), including the subject number and the SVR visit window corresponding to the first occurrence of relapse. A similar listing will be prepared for subjects who prematurely discontinued treatment and relapsed after having HCV RNA < LLOQ at their Final Treatment Visit.

The number and percentage of subjects who do not achieve SVR<sub>12</sub> will be summarized by reason for non-response (as defined in Section 10.1). A listing of subject numbers and reason for non-response will be prepared. A similar summary and listing will be prepared for subjects who do not achieve SVR<sub>24</sub>.

The concordance between  $SVR_{12}$  and  $SVR_{24}$  will be assessed by the agreement between  $SVR_{12}$  and  $SVR_{24}$  and the positive predictive value (PPV) and negative predictive value (NPV) of  $SVR_{12}$  on  $SVR_{24}$ . The agreement between  $SVR_{12}$  and  $SVR_{24}$  is a percentage defined as the number of subjects achieving both  $SVR_{12}$  and  $SVR_{24}$  and the number of subjects where both  $SVR_{12}$  and  $SVR_{24}$  are not achieved. The PPV of  $SVR_{12}$  on  $SVR_{24}$  is the proportion of subjects who achieved  $SVR_{12}$  and  $SVR_{24}$  out of all subjects who achieved  $SVR_{12}$ . The NPV of  $SVR_{12}$  on  $SVR_{24}$  is the proportion of subjects who neither achieve



 $SVR_{12}$  nor  $SVR_{24}$  out of all subjects who did not achieve  $SVR_{12}$ . Similarly, the concordance between  $SVR_4$  and  $SVR_{12}$  will be summarized.

### 10.8 Resistance Analyses

For all subjects, full length NS3/4A or NS5A from baseline samples will be sequenced by next generation sequencing (NGS). For subjects who experience virologic failure (ontreatment virologic failure or post-treatment relapse as defined in Section 10.1), full length NS3/4A and NS5A genes from the first sample after virologic failure with HCV RNA  $\geq$  1000 IU/mL will be sequenced by NGS. An appropriate subtype specific prototypic reference sequence will be used for comparison with sequences from samples. Subjects who experience virologic failure will be referred to as subjects in the primary virologic failure (PVF) population, and a listing by subject that includes HCV subtype, IL28B genotype, reason for SVR<sub>12</sub> non-response, time point(s) sequenced as closest to time of VF, and HCV RNA value at the VF time point(s) will be produced for these subjects. In addition, all listings described below will display HCV subtype and reason for SVR<sub>12</sub> non-response in the subject identifier for each subject. A separate listing will delineate all subjects in the PVF population for whom no sequencing was performed (e.g., lost to follow-up while HCV RNA  $\leq$  1000 IU/mL).

Subjects treated with study drug who do not achieve  $SVR_{12}$  due to reasons other than virologic failure (prematurely discontinued study drug with no on-treatment virologic failure, HCV reinfection, missing  $SVR_{12}$  data or other reasons as described in Section 10.1, Reasons for  $SVR_{12}$  Non-Response), but have a time point with HCV RNA  $\geq 1000$  IU/mL after treatment discontinuation, will have the sample at that time point sequenced. These subjects will be referred to as the non-PVF population. A listing of all subjects in the non-PVF population with post-baseline sequencing available will be created that is similar to the listing of subjects in the PVF population with post-baseline sequencing available.



For each DAA target, resistance-associated signature amino acid positions and a key subset of amino acid are listed in Table 6. Appropriate subtype specific prototypic reference sequence will be used for comparison with sequences from samples.

Table 6. List of Genotype-Specific Signature Amino Acid Positions and a Key Subset of Amino Acid Positions

| Genotype | Signature Amino Acid Positions | Key Subset of Amino Acid Positions |
|---|---|---|
| NS3/4A | | |
| 1a | 36, 43, 54, 55, 56, 80, 107, 122, 132, 155, 156, 158, 168, and 170 | 155, 156, 168 |
| 1b | 36, 54, 55, 56, 80, 107, 122, 155, 156, 158, 168, 170, and 175 | 155, 156, 168 |
| 2, 3, 4, 5, 6 | 36, 43, 54, 55, 56, 80, 155, 156, 166 (GT3 only) and 168 | 155, 156, 168 |
| NS5A | | |
| 1a | 24, 28, 29, 30, 31, 32, 58, 62, 92,<br>and 93 | 24, 28, 30, 31, 58, 92, 93 |
| 1b | 24, 28, 29, 30, 31, 32, 54, 58, 62,<br>92, and 93 | 24, 28, 30, 31, 58, 92, 93 |
| 2, 3, 4, 5, 6 | 24, 28, 29, 30, 31, 32, 58, 92, and 93 | 24, 28, 30, 31, 58, 92, 93 |

Included time points for analyses on samples from subjects who do not achieve  $SVR_{12}$  are 1) the sample closest in time after failure/discontinuation with an HCV RNA level of  $\geq 1000$  IU/mL, and 2) 24 weeks post-DAA treatment, provided that resistance-associated variants were detected at the time of failure/discontinuation

The following definitions will be used in the resistance analyses:

- Baseline variant: a variant by NGS in a baseline sample (≥ 2% or ≥ 15% prevalence within a subject's viral population depending on variant frequency threshold utilized) that was not present in the appropriate prototypic reference amino acid sequence for a given DAA target (NS3/4A or NS5A)
- Variant at signature amino acid position: variant (relative to reference) present by NGS at a detection threshold of  $\geq 2\%$  or  $\geq 15\%$  (depending on variant



- frequency threshold utilized) within a subject's viral population in a baseline or a post-baseline sample at a signature amino acid position
- Post-baseline variant: an amino acid variant in a post-baseline time point sample that was not detected at baseline (< 2%) in the subject and is detectable in ≥ 2% of the sequences from the post-baseline sample
- Enriched variant: variant present in both the baseline and a post-baseline sample whose prevalence in the post-baseline sample is at least 20 percentage points greater than the prevalence in the baseline sample [(post-baseline % − baseline %) ≥ 20]
- Treatment-emergent variant by NGS: A post-baseline variant or an enriched variant

#### Analysis will be Performed Separately for each HCV Subtype Within each Listing.

**Analysis 1:** The following analyses will be performed for all subjects:

- A listing of all baseline variants (≥ 2% detection threshold) at signature resistance-associated amino acid positions for each DAA target (NS3/4A and NS5A) (ITT).
- A listing of all baseline variants (≥ 15% detection threshold) at non-signature resistance-associated amino acid positions for each DAA target (NS3/4A and NS5A) for subjects in PVF population.
- A listing of baseline variants (≥ 15% detection threshold) at signature amino acid positions in subjects with variants across both NS3 and NS5A, or those with multiple baseline variants within any one target (NS3 or NS5A) (ITT population).
- The number and percentage of subjects with baseline variants at detection-thresholds of ≥ 2% and ≥ 15% for variants at signature amino acid positions (ITT). This table includes prevalence of each baseline variant, and a summary of number of subjects with variants in NS3 only, NS5A only, and NS3 + NS5A. Include the number of GT2 − 6 subjects with variants in NS3 only, NS5A only, any in NS3, any in NS5A, any in NS3 or NS5A, any in NS3 + NS5A.



- Total number and percentage of subjects with baseline polymorphisms *at a key subset of amino acid positions* in NS3 only, in NS5A only, any in NS3, any in NS5A, any in NS3 or NS5A, any in NS3 + NS5A (ITT), by subtype, and total.
- Total number and percentage of subjects with baseline polymorphisms *at a key subset of amino acid positions* in NS3 only, in NS5A only, any in NS3, any in NS5A, any in NS5A, any in NS5A, any in NS5A, any in NS5A, any in NS5A (ITT), by genotype, and total.

**Analysis 2:** The impact of baseline variants on treatment outcome will be assessed for **mITT-GT-VF** population as follows: for each variant, the  $SVR_{12}$  rate will be calculated for subjects with and without the variant and the 2 rates will be compared using Fisher's exact test. Analysis will be grouped by HCV subtype and DAA target (NS3/4A or NS5A). The analysis will include total number of subjects within each subtype with any variant within NS3, any variant within NS5A, and with variants in NS3 + NS5A.

The following will be included in the analyses of impact of baseline variants on treatment outcome:

- Variants at signature amino acid positions (vs no variant at that position), using detection thresholds of both 2% and 15%. The analysis will include the number of subjects with variants in NS3 only, in NS5A only, any in NS3, any in NS5A, any in NS3 or NS5A, any in NS3 + NS5A.
- Variants at each non-signature amino acid position at a detection threshold of 15%.
- Each variant at signature amino acid position (vs not that variant) using detection thresholds of 2% and 15%. The analysis will include the number of subjects with variants in NS3 only, in NS5A only, any in NS3, any in NS5A, any in NS3 or NS5A, any in NS3 + NS5A.

**Analysis 3**: In subjects with or without polymorphisms in NS3 only, in NS5A only, any in NS3, any in NS5A, any in NS5A, any in NS5A, any in NS5A at the *key subset of amino acid positions* at 15% detection threshold, the SVR<sub>12</sub> rate will be calculated, and the rates with or without polymorphisms will be compared using Fisher's exact test.



Analysis will be separated by HCV subtype. The following tables will be provided (mITT-GT-VF):

- Comparison of SVR<sub>12</sub> rates by subtype, and total (include all subtypes)
- Comparison of SVR<sub>12</sub> rates by genotype, and total (include all subtypes)

# Analysis 4 (will be available in the primary CSR and will updated in the final CSR for the study):

The following analyses will be performed for subjects who do not achieve SVR<sub>12</sub> (with separate summaries for subjects in PVF and non-PVF populations) and have post-baseline resistance data available:

- Listings by subject of all *treatment-emergent variants* relative to the baseline amino acid sequences will be provided for each DAA target (NS3/4A and NS5A).
- Listings by subject of all *variants at signature amino acid positions* in a post-baseline time point for each DAA target (NS3/4A and NS5A).
- The persistence of post-baseline variants at signature resistance-associated amino acid positions for each target (NS3 and NS5A) from subjects will be assessed at Post-Treatment Week 24. Listings by subject and time point of all treatment-emergent variants will be provided for each DAA target (NS3 and NS5A).

#### **HCV Genotype/Subtype**

Phylogenetic analysis will be conducted on HCV sequence from baseline samples from all subjects in order to accurately determine subtype.

Subjects' HCV genotype and subtype may be assessed based on the Inno-LiPA 2.0 Assay used by the Central lab (Covance), the HCV genotype determination by Sanger sequencing a region of NS5B by the Central lab (Covance) and/or from phylogenetic analysis of the full length NS3/4A, and/or NS5A sequences performed by AbbVie. If the


ABT-493/ABT-530 M13-596 – Statistical Analysis Plan Version 1.0 – 27 October 2016

phylogenetic analysis is available, then it will be used to determine the subject's HCV genotype and subtype. If it is not available, then the Sanger sequencing assay result will be used to determine the subject's HCV genotype and subtype, if available. Finally, if neither the phylogenetic analysis result nor the Sanger sequencing assay results is available, then the Inno-LIPA assay results will be used to categorize the subject. This subtype information will be presented in summaries of efficacy subgroup analyses. The baseline characteristic summary will use the results from the central laboratory (Sanger sequencing or Inno-LiPA 2.0 Assay [if Sanger sequencing not available]).

This subtype information will be presented in summaries of efficacy subgroup analyses. The baseline characteristic summary will use the results from the central laboratory (Sanger sequencing or Inno-LiPA 2.0 Assay [if Sanger sequencing not available]).

A summary of HCV subtype as provided by the central laboratory (Sanger sequencing or Inno-LiPA 2.0 Assay [if Sanger sequencing not available]) versus phylogenetic analysis also will be provided.

#### 10.8.1 Presence of Baseline Resistance-Associated Variants

For the efficacy subgroup analyses defined in Section 10.6, any NS3/4A variant and any NS5A variant are defined as follows, where baseline resistance-associated variants based on  $\geq$  15% NGS detection threshold are considered. Signature amino acid positions of NS3/4A and NS5A by HCV genotype are listed in Table 7.



Table 7. Resistance-Associated Variants by DAA Target and HCV Genotype

| Target | Genotype | Signature Amino Acid Positions<br>(All Variants at These<br>Positions Are to Be Included) | Other Specific Variants |
|---|---|---|---|
| NS3/4A | 1, 2, 3, 4, 5, 6 | 155, 156, 168 | |
| NS5A | 1a | 28, 30, 31, 93 | H58D, E62A |
| | 1b | 31, 93 | |
| | 2 | 24, 28, 30, 92, and 93 | |
| | 3 | 24, 28, 30, 31, 58, and 93 | |
| | 4 | 24, 28, 30, 31, and 93 | |
| | 5 | 24, 28, 30, 31, 58, 92, and 93 | |
| | 6 | 24, 28, 30, 31, 58, 92, and 93 | |

For example, according to Table 7, all subjects with any baseline variant at amino acid positions 155, 156, or 168 will be counted as having any NS3/4A variant at baseline; any HCV genotype 2 subjects with any baseline variant at amino acid positions 24, 28, 30, 92, or 93 will be counted as having any NS5A variant at baseline.

The number and percent of subjects in the mITT-GT-VF population will be summarized for the presence of baseline resistance-associated variants of:

- 1. Any NS3/4A variant at baseline (yes/no);
- 2. Any NS5A variant at baseline (yes/no);
- 3. Any NS3/4A variant at baseline or any NS5A variant at baseline (yes/no);
- 4. Both NS3/4A and NS5A variant at baseline (i.e., any NS3/4A variant at baseline and any NS5A variant at baseline) (yes/no);
- 5. Presence or absence of any variant
  - 5a. Any NS3/4A variant at baseline only (i.e., without baseline NS5A variants);
  - 5b. Any NS5A variant at baseline only (i.e., without baseline NS3/4A variants);
  - 5c. Both NS3/4A and NS4A variant at baseline;

5d. None (i.e., no baseline variant in either NS3/4A or in NS5A at baseline).

## 10.9 Patient Reported Outcomes

The following instruments will be used to collect patient reported outcomes (PROs): SF-36 version 2 (SF-36v2), Fatigue Severity Scale (FSS), and EuroQol-5 Dimensions-3 Level (EQ-5D-3L).

Subject's responses to the EQ-5D-3L will be combined into a unique health state using a 5-digit code with 1 digit from each of the 5 dimensions. The EQ-5D-3L states will be converted into a single preference-weighted health utility index score by applying weights.<sup>1,2</sup> The VAS score will be analyzed separately.

The SF-36v2 measures dimensions of a patient's functional health and well-being in 8 domains and also provides 2 summary scores that characterize a patient's mental (Mental Component Summary; MCS) and physical (Physical Component Summary; PCS) health status. Imputation will be applied to each domain as described in Section 6.3. The score for each of the 8 domains ranges from 0 to 100 and will be normalized according to the user manual. The standardization of the normalized scores will provide the norm-based scores with a mean of 50 and a SD of 10. The two summary scores are based on the norm-based scores. Per the SF-36v2 instrument manual, score for any item with multiple responses will be set to "missing." Subject's responses to the SF-36v2 will be summarized for the PCS and MCS measures and eight individual domain measures.

The FSS measures the impact of fatigue over the past week on specific types of functioning. The survey consists of 9 questions using a 7-point Likert scale. A total score is calculated as the average of the individual item responses (adding up all the answers and dividing by nine). Higher FSS scores indicate a higher degree of impact of fatigue. Imputation will be applied to the total score as described in Section 6.3.

Summary statistics (n and mean) at each visit and for change from baseline (n, mean, SD, minimum and maximum) to each visit will be provided for the SF-36v2 (MCS and PCS)



abbvie ABT-493/ABT-530 M13-596 – Statistical Analysis Plan Version 1.0 – 27 October 2016

scores; FSS total score; and EQ-5D-3L health index score and VAS score and will be summarized descriptively at each visit and for change from baseline to each visit.

The following analyses of patient reported outcomes (PROs) also will be performed:

- Number and percentage of subjects who have ever experienced an increase from baseline up through each applicable time point of greater than or equal to 2.5 points in the SF-36 MCS and PCS, along with two-sided 95% Normal CI;
- Number and percentage of subjects who have ever experienced an increase from baseline up through each applicable time point of greater than or equal to 5 points in the SF-36 domain scores, along with two-sided 95% Normal CI;
- Number and percentage of subjects who have ever experienced an increase from baseline up through each applicable time point of greater than or equal to 0.7 in the FSS total score, along with two-sided 95% Normal CI.

If a subject starts another treatment for HCV, then all PRO values for this subject measured on or after the start date of the new HCV treatment will be excluded from analyses.

#### 11.0 **Safety Analysis**

#### 11.1 **General Considerations**

Safety data will be summarized using the safety population.

#### 11.2 **Analysis of Adverse Events**

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The actual version of the MedDRA coding dictionary will be noted in the clinical study report.

#### 11.2.1 **Treatment-Emergent Adverse Events**

Treatment-emergent adverse events are defined as any adverse event (AE) with an onset date that is after the first dose of study drug and no more than 30 days after the last dose of study drug. Events where the onset date is the same as the study drug start date are



assumed to be treatment-emergent. If an incomplete onset date was collected for an adverse event, the event will be assumed to be treatment-emergent, unless there is other evidence that confirms that the event was not treatment-emergent (e.g., the event end date was prior to the study drug start date).

## 11.2.2 Tabulations of Treatment-Emergent Adverse Events

The number and percentage of subjects will be tabulated by primary MedDRA System Organ Class (SOC) and preferred term (PT). The system organ classes will be presented in alphabetical order, and the preferred terms will be presented in alphabetical order within each system organ class.

#### **Adverse Event Overview**

An overview of AEs will be presented consisting of the number and percentage of subjects experiencing at least one event for each of the following AE categories:

- Any treatment-emergent adverse event;
- Treatment-emergent adverse events with a "reasonable possibility" of being related to DAAs (ABT-493/ABT-530);
- Treatment-emergent adverse events of Grade 3 or higher;
- Serious treatment-emergent adverse events;
- Serious treatment-emergent adverse events with a "reasonable possibility" of being related to DAAs (ABT-493/ABT-530);
- Treatment-emergent adverse events leading to discontinuation of study drug;
- DAA-related treatment-emergent adverse events leading to discontinuation of study drug;
- Treatment-emergent adverse events of Grade 3 or higher with a "reasonable possibility" of being related to DAA (ABT-493/ABT-530);
- Serious treatment-emergent adverse events leading to discontinuation of study drug;
- Treatment-emergent adverse events leading to interruption of study drug;
- Treatment-emergent adverse events leading to death;



• Deaths.

## **Adverse Events by SOC and PT**

Subjects reporting more than one AE for a given PT will be counted only once for that term (most severe/highest grade incident for the severity tables and most related incident for the relationship tables). Subjects reporting more than one AE within an SOC will be counted only once for that SOC. Subjects reporting more than one AE will be counted only once in the overall total.

The following summaries of AEs by SOC and PT will be generated:

- Treatment-emergent adverse events;
- Treatment-emergent adverse events with a "reasonable possibility" of being related to DAAs (ABT-493/ABT-530);
- Serious treatment-emergent adverse events;
- Serious treatment-emergent adverse events with a "reasonable possibility" of being related to DAAs (ABT-493/ABT-530);
- Grade 3 or higher treatment-emergent adverse events;
- Treatment-emergent adverse events of Grade 3 or higher with a "reasonable possibility" of being related to DAAs (ABT-493/ABT-530);
- Treatment-emergent adverse events leading to discontinuation of study drug;
- DAA-related treatment-emergent adverse events leading to discontinuation of study drug;
- Serious treatment-emergent adverse events leading to discontinuation of study drug;
- Treatment-emergent adverse events leading to interruption of study drug;
- Treatment-emergent adverse events leading to death.

A listing of treatment-emergent adverse events grouped by body system and preferred term with subject numbers will be created.



abbvie ABT-493/ABT-530 M13-596 - Statistical Analysis Plan Version 1.0 – 27 October 2016

#### **Adverse Events by PT**

The number and percentage of subjects experiencing treatment-emergent adverse events will be tabulated according to PT and sorted by overall frequency. Similar summaries will be provided for Grade 3 or higher treatment-emergent adverse events, DAA-related treatment-emergent adverse events, DAA-related Grade 3 or higher treatment-emergent adverse events, and DAA-related treatment-emergent serious adverse events.

#### **Adverse Events by Maximum Severity Grade Level**

Treatment-emergent adverse events and DAA-related treatment-emergent adverse events will be summarized by maximum severity grade level of each preferred term. Each adverse event will be assigned a grade level (Grade 1, 2, 3, 4, or 5) by the investigator. If a subject has an AE with unknown severity, then the subject will be counted in the severity grade level category of "unknown," even if the subject has another occurrence of the same event with a severity present. The only exception is if the subject has another occurrence of the same AE with the highest grade level (Grade 5). In this case, the subject will be counted under the "Grade 5" category.

#### **Adverse Event by Maximum Relationship**

Treatment-emergent adverse events also will be summarized by maximum relationship of each preferred term to study drug (DAA), as assessed by the investigator. If a subject has an adverse event with unknown relationship, then the subject will be counted in the relationship category of "unknown," even if the subject has another occurrence of the same event with a relationship present. The only exception is if the subject has another occurrence of the same adverse event with a relationship assessment of "Reasonable Possibility." In this case, the subject will be counted under the "Reasonable Possibility" category.

#### **Other Adverse Events**

The number and percentage of subjects experiencing at least one treatment-emergent adverse event in the search defined below by Product MedDRA Query (PMQ) will be



presented overall and by SOC and PT. In addition, a listing of treatment-emergent adverse events for subjects meeting the search criterion will be provided.

"Hepatic Decompensation and Hepatic Failure" (PMQ)

#### 11.2.3 Listing of Adverse Events

The following listings of adverse events will be prepared:

- All serious adverse events (from the time the subject signed the study-specific informed consent through the end of the study),
- Treatment-emergent serious adverse events,
- Treatment-emergent adverse events leading to death,
- Treatment-emergent adverse events leading to discontinuation of study drug,
- Treatment-emergent adverse events leading to study drug interruption.

# 11.3 Analysis of Laboratory Data

Data collected from the central and local laboratories, including additional laboratory testing due to an SAE, will be used in all analyses.

## 11.3.1 Variables and Criteria Defining Abnormality

Hematology variables include: hematocrit, hemoglobin, red blood cell (RBC) count, white blood cell (WBC) count, neutrophils, bands, lymphocytes, monocytes, basophils, eosinophils, platelet count, reticulocyte count, prothrombin time (PT), international normalized ratio (INR), and activated partial thromboplastin time (aPTT).

Chemistry variables include: blood urea nitrogen (BUN), creatinine, total bilirubin, direct and indirect bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, sodium, potassium, calcium, inorganic phosphorus, cholesterol, total protein, glucose, triglycerides, albumin, chloride, bicarbonate, magnesium, total insulin, gamma-glutamyl transferase (GGT), creatinine clearance (calculated using

Cockcroft-Gault), and estimated glomerular filtration rate (eGFR) calculated using the modification of diet in renal disease (MDRD) equation defined below.

Urinalysis variables include: specific gravity, ketones, pH, protein, blood, glucose, urobilinogen, bilirubin, leukocyte esterase, and microscopic (reflexly performed if other variables are abnormal).

Some of the above laboratory variables are calculated by the laboratory vendor including indirect bilirubin, creatinine clearance, and eGFR by MDRD. The central lab calculates eGFR by MDRD using the following equation, where serum creatinine is measured in mg/dL and age is measured in years:

The central lab calculates the estimated creatinine clearance (CrCl) based on the following Cockcroft-Gault formula:

CrCl (mL/min) = 
$$[(140 - age) \times (weight in kg) \times (0.85 if female)]/[serum creatinine (mg/dL) \times 72].$$

#### 11.3.2 Statistical Methods

The baseline value for clinical laboratory tests will be the last non-missing measurement on or before the day of the first dose of study drug. Values on Day 1 must also be before the time of first dose if time is available. The same baseline value will be used for change to Treatment Period visits and change to Post-Treatment Period visits.

Mean changes from baseline to each post-baseline visit, including applicable post-treatment visits, will be summarized. Each protocol-specified laboratory parameter will be summarized with the sample size, baseline mean, visit mean, change from baseline mean, standard deviation, minimum, median, and maximum.

The laboratory parameters defined in Table 8 will be assigned a toxicity grade of 1, 2, 3, or 4. The number and percentage of subjects with a maximum toxicity grade of 1, 2, 3 or 4, will be summarized. The post-baseline value must be in a toxicity grade that is more extreme than the toxicity grade corresponding to the baseline value to be counted. The summary will also include the number and percentage of subjects with a maximum of at least Grade 3 for all laboratory parameters in Table 8. A listing of all relevant laboratory parameters will be provided for each subject who had an increase to Grade 2 or higher for all laboratory variables in Table 8.

Table 8. Definitions of Toxicity Grades 1, 2, 3, and 4 for Laboratory Values

| Test | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| ALT/SGPT | $>$ ULN $-3 \times$ ULN | $> 3 - 5 \times ULN$ | $> 5 - 20 \times ULN$ | > 20 × ULN |
| AST/SGOT | $>$ ULN $-3 \times$ ULN | $> 3 - 5 \times ULN$ | $> 5 - 20 \times ULN$ | $> 20 \times ULN$ |
| Alkaline Phosphatase | $>$ ULN $-2.5 \times$ ULN | $> 2.5 - 5 \times ULN$ | $> 5 - 20 \times ULN$ | $> 20 \times ULN$ |
| Total Bilirubin | $>$ ULN $-$ 1.5 $\times$ ULN | $> 1.5 - 3 \times ULN$ | $> 3 - 10 \times ULN$ | $> 10 \times ULN$ |
| Hemoglobin | < LLN $-$ 100 g/L | < 100 - 80 g/L | < 80 g/L | |
| Absolute Neutrophil<br>Count | $< LLN - 1.5 \times 10^9 / L$ | $< 1.5 - 1.0 \times 10^9 / L$ | $< 1.0 - 0.5 \times 10^9 / L$ | $<0.5\times10^9/L$ |
| Platelet count | $<$ LLN $-75.0 \times 10^9$ /L | $< 75.0 - 50.0 \times 10^9 / L$ | $< 50.0 - 25.0 \times 10^9 / L$ | $< 25.0 \times 10^9 / L$ |
| INR | $> 1 - 1.5 \times ULN$ | $> 1.5 - 2.5 \times ULN$ | > 2.5 × ULN | |
| Creatinine clearance | < LLN $-$ 60 mL/min | < 60 – 30 mL/min | < 30 – 15 mL/min | < 15 mL/min |
| Creatinine | $>$ ULN $-$ 1.5 $\times$ ULN | $> 1.5 - 3 \times ULN$ | $> 3 - 6 \times ULN$ | $> 6 \times ULN$ |
| Albumin | < LLN $-30$ g/dL | < 30 - 20 g/L | < 20 g/L | |

#### **Assessment of Hepatic Laboratory Parameters**

The number and percentage of subjects with maximum on-treatment lab values meeting the following criteria will be summarized:

- ALT  $\geq$  3 × ULN and total bilirubin  $\geq$  2 × ULN;
- ALT  $\geq$  3 × ULN and total bilirubin < 2 × ULN;
  - $\circ$  ALT > 5 × ULN and total bilirubin < 2 × ULN;
- ALT  $< 3 \times$  ULN and total bilirubin  $\ge 2 \times$  ULN.



The maximum ratio relative to the ULN will be used to determine if subjects meet the criteria listed above. The ALT and total bilirubin values do not need to be concurrent in order to meet the defined criteria. For ALT, the post-baseline value must represent an increase from the first nadir (including baseline) to be counted. First nadir is defined as the last value prior to the first increase. For total bilirubin, a subject will be counted if the post-baseline laboratory value meets the above criteria regardless of the baseline laboratory value (i.e., the post-baseline laboratory value does not need to be worse than the baseline laboratory value).

A listing of all ALT, AST, total, indirect and direct bilirubin, ratio of direct to total bilirubin, and alkaline phosphatase values will be provided for each subject who met any of the criteria defined above. The listings will be reviewed to assess bilirubin (e.g., mixed or direct predominance) and temporal relationships for subjects with ALT  $\geq$  3 × ULN and total bilirubin  $\geq$  2 × ULN.

The number and percentage of subjects with post-baseline values during the Treatment Period meeting the following criteria will be summarized:

- ALT  $> 5 \times ULN$  and  $\geq 2 \times baseline$ ;
- AST  $> 5 \times ULN$  and  $\geq 2 \times baseline$ ;
- Total bilirubin  $\geq 2.0 \times ULN$  and > baseline.

As noted above, a post-baseline value must be more extreme than the baseline value to be considered. A separate listing will be provided that presents all lab values for the subjects meeting any of these criteria during treatment.

#### 11.4 Analysis of Vital Signs and Weight

## 11.4.1 Variables and Criteria Defining Abnormality

Vital sign variables are body temperature, sitting systolic blood pressure, sitting diastolic blood pressure, sitting pulse rate, and body weight.



The criteria for potentially clinically significant vital sign findings are presented in Table 9.

Table 9. Criteria for Potentially Clinically Significant Vital Sign Values

| Test/Measurement | Very Low (VL) | Very High (VH) |
|---|---|---|
| Systolic Blood Pressure | $\leq$ 90 mmHg AND A decrease of $\geq$ 20 mmHg from baseline | ≥ 180 mmHg AND An increase of ≥ 20 mmHg from baseline |
| Diastolic Blood Pressure | $\leq$ 50 mmHg AND A decrease of $\geq$ 15 mmHg from baseline | ≥ 105 mmHg AND An increase of ≥ 15 mmHg from baseline |
| Pulse Rate | ≤ 50 bpm AND A decrease of ≥ 15 bpm from baseline | ≥ 120 bpm AND An increase of ≥ 15 bpm from baseline |
| Weight | A decrease of ≥ 15% from baseline | An increase of $\geq$ 15% from baseline |
| Body Temperature | | > 38.3°C AND An increase of<br>≥ 1.1°C from baseline |

#### 11.4.2 Statistical Methods

The baseline value for vital signs will be the last measurement on or before the day of the first dose of study drug. The same baseline value will be used for change to Treatment Period visits and change to Post-Treatment Period visits.

Mean changes from baseline to each post-baseline visit, including applicable post treatment visits, will be summarized. Each vital sign parameter will be summarized with the baseline mean, visit mean, change from baseline mean, standard deviation, minimum, median, and maximum.

The number and percentage of subjects with on-treatment values meeting the specified criteria for Potentially Clinically Significant (PCS) vital sign values (Table 9) will be summarized. A post-baseline value must be more extreme than the baseline value to be considered a PCS finding. A separate listing will be provided that presents all vital sign values for the subjects meeting PCS criteria during treatment.



M13-596 – Statistical Analysis Plan Version 1.0 – 27 October 2016

# 12.0 Summary of Changes

# 12.1 Summary of Changes Between the Latest Version of Protocol and SAP

- 1. Updates were made to the resistance analysis plan to be consistent across the HCV ABT-493/ABT-530 program.
- 2. Updates were made to the subgroup efficacy analysis section to be consistent across the HCV ABT-493/ABT-530 program

## 13.0 References

- 1. Szende A, Williams A. Measuring self-reported population health: an international perspective based on EQ-5D. EuroQol Group Monographs Volume 1. SpringMed Publishing; 2004.
- 2. Rabin R, Oemar M, Oppe M, et al. EQ-5D-5L user guide: basic information on how to use the EQ-5D-5L instrument, Version 1.0. Rotterdam, the Netherlands: EuroQol Group; 2011.
- 3. Ware JE Jr, Kosinski M, Bjorner JB, et al. User's manual for the SF-36v2 health survey. 2nd ed. Lincoln, RI: QualityMetric Incorporated; 2007.

# **Document Approval**

Study M13596 - Statistical Analysis Plan Version 1 - 27Oct2016 (E3 16.1.9)

Version: 1.0 Date: 27-Oct-2016 08:34:39 PM Company ID: 10272016-00F9F681391D61-00001-en

| Signed by: | Date: | Meaning Of Signature: |
|------------|-------------------------|-----------------------|
| | 27-Oct-2016 03:18:41 PM | Author |
| | 27-Oct-2016 04:15:50 PM | Approver |
| | 27-Oct-2016 07:38:56 PM | Approver |
| | 27-Oct-2016 08:34:34 PM | Approver |